CLINICAL TRIAL: NCT02639624
Title: Altering Bicarbonate Delivery During Hemodialysis to Affect Filtration of Indoxyl Sulfate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: 07/27/2017 Unable to contact research team to confirm reason for withdrawing study.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-01343
Record Dates: First submitted 2015-12-22; First posted 2015-12-24 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Renal Dialysis; Hemodialysis
Keywords: hemodialysis; kidney; dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low bicarbonate dialysate First (Experimental): Dialysis with low bicarbonate dialysate (expected normal for an adult ~24 mEq) for the first half of dialysis then switched over to normal bicarbonate dialysate for the second half.
  Interventions: Drug: Low bicarbonate dialysate First; Drug: Normal bicarbonate dialysate
- Normal bicarbonate dialysate First (Active Comparator): Dialysis with normal (37 mEq) for the first half of dialysis then switched over to low bicarbonate dialysate
  Interventions: Drug: Normal bicarbonate dialysate First; Drug: Low bicarbonate dialysate

INTERVENTIONS:
Drug: Low bicarbonate dialysate First
  Arms: Low bicarbonate dialysate First
Drug: Normal bicarbonate dialysate First
  Arms: Normal bicarbonate dialysate First
Drug: Normal bicarbonate dialysate
  Arms: Low bicarbonate dialysate First
Drug: Low bicarbonate dialysate
  Arms: Normal bicarbonate dialysate First

SUMMARY:
This is a non randomized crossover trial investigating whether changing the pattern of bicarbonate administration during hemodialysis will result in the more efficient filtration of highly protein bound solutes. The experimental group will be dialyzed with low bicarbonate dialysate for the first half of dialysis then switched over to normal bicarbonate dialysate for the second half. The control group will be dialyzed entirely with normal bicarbonate dialysate. The two groups will switch one week late and patients will serve as their own matched controls for a completely standard dialysis and one that is split into two halves with different bicarbonate concentrations.

DETAILED DESCRIPTION:
Investigators will try to perform dialysis with a low bicarbonate bath which will leave patients blood pH (Hydrogen ion concentration) relatively unchanged then switch to a normal bicarbonate bath during the second half of dialysis so that they attain the pH (Hydrogen ion concentration) they normally would. Investigators will use these measurements to test test the hypothesis that Indoxyl Sulfate (IS) binds to proteins with greater affinity under basic conditions and further to test the hypothesis that it is possible to remove a greater amount of Indoxyl Sulfate (IS) when patients are maintained relatively acidotic during dialysis for a longer period of time due to the greater availability of free IS that can pass through the dialyzer.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Stable Dialysis for at least 6 months

Exclusion Criteria:

* Patients with serum potassium concentration below 4.0 mEq/L on previous monthly lab test or corrected serum calcium below 8.5 mEq/L
* Hospitalization within the past 12 months
* Adults unable to consent
* Children
* Pregnant women
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change in the amount of Indoxyl Sulfate level in the first half of dialysis as compared to controls | 1 Minute, 75 Minutes, 105 Minutes, 180 Minutes, 210 Minutes

SECONDARY OUTCOMES:
Change in pH | 1 Minute, 75 Minutes, 105 Minutes, 180 Minutes, 210 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Lowenstein, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States